CLINICAL TRIAL: NCT02739503
Title: Fetal Head Circumference as a Predictor of Operative Delivery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0017-16-HYMC
Record Dates: First submitted 2016-04-07; First posted 2016-04-15 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Pregnancy
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Ultrasound — Patients will receive ultrasound in the ultrasound unit at Hillel Yaffe Medical Center within 10 days before onset of induced or spontaneous labors. The ultrasound team has been trained in FHC , Estimated Fetal Weight (EFW) and Biparietal Diameter (BPD) measurement .Optimal ultrasound measurements of FHC and BPD will be obtained. The average of 3 fetal head circumference measurements will be recorded. Investigators consider the FHC and BPD to be optimal when a clear outline of the entire fetal skull is measured, and the landmarks (the thalamus, cavum septum pellucidum and choroid plexus in the atrium of the lateral ventricles) are visualized. Subsequent information of labor outcome as well as normal head circumference ,post-delivery will be obtained from maternal and neonatal medical records.

SUMMARY:
This study set out to investigate whether antenatal ultrasound evaluation of the Fetal Head Circumference (FHC) could potentially possess a predictive role in determining women at increased risk for operative delivery or cesarean section.

DETAILED DESCRIPTION:
When vaginal delivery poses a danger to the mother or newborn infant, operative delivery (instrumental or cesarean section) is indicated. Some specific indications for operative delivery include prolonged second-stage of labor, suspected compromise of the fetus, health-related disorders of the fetus or the mother that justify shortening of the second-stage of active labor and more. In cases where cephalo-pelvic disproportion (CPD) is suspected or when instrumental delivery is not possible or fails, cesarean section plays a critical role . Studies trying to identify women at greatest risk of CPD have concluded that neither x ray, nor computed tomography or magnetic resonance imaging have a proven value in labor management or in predicting clinical outcomes . Previous studies assessing fetal factors that are associated with operative delivery have focused mainly on estimated fetal weight to predict macrosomia. Nonetheless, ultrasound estimation of the fetal weight was shown to differ by as much as 20% from actual birth weight, and identifying cases with suspected fetal macrosomia, other than for diabetic pregnancies, was not found to improve labor outcome . As weeks may possibly elapse between the time of last antenatal assessment and onset of labor, a further challenge is related to the timing of ultrasound assessment. Several studies have shown an association between increased Fetal Head Circumference (FHC) and prolonged second-stage of labor, instrumental delivery and cesarean section . However, FHC can only be acquired following delivery and has no predictive value for interventions in labor.

ELIGIBILITY:
Inclusion Criteria:

1. Women at term (37+0 - 42+0 weeks' gestation)
2. Singleton pregnancies
3. Cephalic presentation
4. Anticipated vaginal delivery

Exclusion Criteria:

1. Younger than 18 years old and older than 45 years old
2. Women who incapable of providing informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women at term (37+0 - 42+0 weeks' gestation)
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The rate of "operative delivery" including instrumental deliveries or cesarean sections. | 1 year

SECONDARY OUTCOMES:
Length (in hours) of the first and second stages of labor. | 1 year
Rate of obstetric anal sphincter injury. | 1 year
Rate of early postpartum hemorrhage (PPH). | 1 year
Rate of neonatal trauma. | 1 year
Rate of admission to the neonatal intensive care unit. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Limonad, M.D, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Department of Obstetrics and Gynecology, Hillel-Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ACOG Practice Bulletin No. 154: Operative Vaginal Delivery. Obstet Gynecol. 2015 Nov;126(5):e56-e65. doi: 10.1097/AOG.0000000000001147. No abstract available. PMID 26488523
- [Background] Murphy DJ, Liebling RE, Verity L, Swingler R, Patel R. Early maternal and neonatal morbidity associated with operative delivery in second stage of labour: a cohort study. Lancet. 2001 Oct 13;358(9289):1203-7. doi: 10.1016/S0140-6736(01)06341-3. PMID 11675055
- [Background] Maharaj D. Assessing cephalopelvic disproportion: back to the basics. Obstet Gynecol Surv. 2010 Jun;65(6):387-95. doi: 10.1097/OGX.0b013e3181ecdf0c. PMID 20633305
- [Background] Lenhard MS, Johnson TR, Weckbach S, Nikolaou K, Friese K, Hasbargen U. Pelvimetry revisited: analyzing cephalopelvic disproportion. Eur J Radiol. 2010 Jun;74(3):e107-11. doi: 10.1016/j.ejrad.2009.04.042. Epub 2009 May 13. PMID 19443160
- [Background] Peregrine E, O'Brien P, Jauniaux E. Clinical and ultrasound estimation of birth weight prior to induction of labor at term. Ultrasound Obstet Gynecol. 2007 Mar;29(3):304-9. doi: 10.1002/uog.3949. PMID 17290365
- [Background] Irion O, Boulvain M. Induction of labour for suspected fetal macrosomia. Cochrane Database Syst Rev. 2000;(2):CD000938. doi: 10.1002/14651858.CD000938. PMID 10796221
- [Background] Elvander C, Hogberg U, Ekeus C. The influence of fetal head circumference on labor outcome: a population-based register study. Acta Obstet Gynecol Scand. 2012 Apr;91(4):470-5. doi: 10.1111/j.1600-0412.2012.01358.x. Epub 2012 Feb 28. PMID 22229662
- [Background] Mujugira A, Osoti A, Deya R, Hawes SE, Phipps AI. Fetal head circumference, operative delivery, and fetal outcomes: a multi-ethnic population-based cohort study. BMC Pregnancy Childbirth. 2013 May 7;13:106. doi: 10.1186/1471-2393-13-106. PMID 23651454
- [Background] Verburg BO, Steegers EA, De Ridder M, Snijders RJ, Smith E, Hofman A, Moll HA, Jaddoe VW, Witteman JC. New charts for ultrasound dating of pregnancy and assessment of fetal growth: longitudinal data from a population-based cohort study. Ultrasound Obstet Gynecol. 2008 Apr;31(4):388-96. doi: 10.1002/uog.5225. PMID 18348183